CLINICAL TRIAL: NCT03751709
Title: IIT2017-05-MERIN-BLINHMCT: Blinatumomab Plus HLA-Mismatched Cellular Therapy (HMCT) for Relapsed/Refractory CD19+ ALL
Brief Title: Blinatumomab Plus HLA-Mismatched Cellular Therapy for Relapsed/Refractory CD19+ ALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Noah Merin, Assistant Clinical Professor, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2017-05-MERIN-BLINHMCT
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: B-Cell Acute Lymphoblastic Leukaemia; ALL, Adult; B-ALL
Keywords: Haplo-Mismatched Cellular Therapy; Acute Lymphoblastic Leukemia; ALL; B-ALL; donor lymphocyte; DLI; blinatumomab; bispecific; microtransplantation; microtransplant
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subjects (Experimental): Blinatumomab+Haplo-Mismatched Cell Therapy (HMCT)
  Interventions: Drug: Blinatumomab; Other: Haplo-Mismatched Cell Therapy (HMCT)

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab per package insert - via continuous infusion days 1-28 of Cycle 1 and Cycle 2, every 42 days.
  Other Names: Blincyto
Other: Haplo-Mismatched Cell Therapy (HMCT) — HMCT infusion Cycle 1, Day 15 and Cycle 2, Day 8 & Day 15
  Other Names: HMCT; 'primary DLI; 'microtransplantation'

SUMMARY:
Single center Phase 1 dose escalation trial of the combination of standard-of-care blinatumomab plus Haplo-Mismatched Cellular Therapy (HMCT). HMCT refers to the infusion of donor peripheral blood mononuclear cells collected via pheresis from a haploidentical family member - the procedure is analogous to giving a donor lymphocyte infusion outside of the setting of an allogeneic stem cell transplant; also known as 'microtransplantation'. The HMCT is an unselected mix of lymphocytes and leukocytes, but the product dose escalation will be done based on the T cell content.

Ten recipients are planned. Each subject will be administered one infusion of HMCT during the first cycle of blinatumomab and two infusions during cycle two of blinatumomab; the CD3+ cell dose of the HMCT infusion is governed by dose escalation / de-escalation following a Bayesian method.

DETAILED DESCRIPTION:
This single center, phase 1 study will examine the safety, side effects, and effectiveness of combining the investigational use of Haplo-Mismatched Cellular Therapy (HMCT) in combination with blinatumomab. Investigators plan to give HMCT starting on day 15, after the initial CRS caused by blinatumomab has resolved. The investigational treatment will start with 1% of the typical HMCT dose (10e6 CD3+ cells/kg) and will employ a modified dose escalation design as an additional safety measure. The primary end points will be DLT of the combination of blinatumomab and HMCT.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/Refractory CD19+ Acute Lymphoblastic Leukemia. Patients with minimal residual disease detected by NGS > 10e-6 or multiparameter flow cytometry > 10e-5 in blood or bone marrow are eligible.
* Patients must belong to one of the following 'high risk' categories: (i) at least 2nd relapse or refractory to at least one salvage therapy (ii) relapse after autologous stem cell transplantation, (iii) any relapse in a patient with no immediate allogeneic transplant option (such as advanced age, comorbidity, lack of identified donor, or patient refusal) (iv) Patients with Ph+ ALL will be allowed on the trial at the discretion of the treating physician if they are no longer candidates for further TKI based therapy. Prior therapy with a minimum of 2 prior 2nd/3rd generation TKI is required. (TKI therapy is not allowed while on trial).
* Patients with prior blinatumomab treatment are eligible if last treatment was at least 3 months prior to C1D1, patient's blasts are confirmed to express CD19, and patient did not develop Grade 4 toxicities with prior blinatumomab therapy.
* Age ≥ 18 years.
* Patient has at least one medically fit first- or second-degree family member who is a potential haploidentical donor. In addition, the prospective donor is willing to voluntarily donate peripheral blood cells, and sign consent forms. For minors, consent will be obtained from parent/guardian (assent from the minor is required).
* Patients must have adequate organ function as defined below (note there are no marrow function criteria, cytopenias will not result in exclusion):

  * Serum creatinine ≤ 2.0 x the upper limits of institutional normal (ULN)
  * Total bilirubin ≤ 1.5x the upper limits of institutional normal, unless elevated bilirubin is attributed to liver involvement of leukemia or Gilbert's disease.
  * AST/ALT ≤ 2.5 x the upper limits of institutional normal (≤ 5 x ULN for patients with suspected liver involvement of leukemia).
* ECOG performance status of 0, 1, or 2, and estimated survival of at least 3 months.
* Patients must be able to understand and agree to sign an IRB-approved informed consent form.
* The effects of treatment on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or complete abstinence) prior to study entry, for the duration of study, and for two months after study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Prior allogeneic stem cell transplant
* Prior treatment with fludarabine or cladribine within the last six months prior to C1D1, or treatment with antithymocyte globulin (ATG) or alemtuzumab within the last 1 year.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or lactating.
* Who have had non-biopsy surgery in the last 10 days.
* Who have active CNS disease. Patients with previously treated leptomeningeal disease without evidence of remaining leukemia cells by spinal fluid will be eligible. Intrathecal chemo may be given for prophylaxis for patients who previously had CNS involvement but have now cleared the CSF, at the discretion of the treating physician. Recommend to avoid IT chemotherapy for a few days before or after HMCT infusion.
* History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis (patients with minor prior stroke who are cognitively intact and capable of performing all ADLs are permitted).
* Patients with known active autoimmune disorder.
* Known infection with HIV virus.
* Patients concurrently taking the following drugs are excluded: mycophenolate, cyclosporine, prednisone > 20mg/day, or immunosuppressive agents (low dose maintenance chemotherapy - POMP, hydroxyurea, low dose prednisone - is allowed until 24 hours prior to starting blinatumomab).
* Patients known to have active hepatitis B or C (Hepatitis B positive patients are allowed if they are on appropriate antiviral agents such as lamivudine).
* Subject likely to not be available to complete all protocol-required study visits or procedures, including follow-up visits, and/or to comply with all required study procedures to the best of the subject and Investigator's knowledge.

History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs | up to 6 months
  Number of Dose Limiting Toxicities experienced by patients undergoing HLA mismatched cellular therapy (HMCT) of allogenic CD3+ cells in combination with blinatumomab.

SECONDARY OUTCOMES:
Number of participants experiencing complete response (CR) from time of transplant to one day following the second treatment | up to 3 months
  Bone marrow aspiration and local peripheral blood counts will be used to measure response. CR is defined as the following:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of disease, AND
  * Full recovery of peripheral blood counts: platelets > 100,000/ul, and ANC > 1000/ul
Number of participants experiencing complete response with partial recovery of peripheral blood counts (CRh) from time of transplant to one day following the second treatment | up to 3 months
  Bone marrow aspiration and local peripheral blood counts will be used to measure response. CRh is defined as the following:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of disease, AND
  * Full recovery of peripheral blood counts: platelets > 50,000/ul, and ANC > 500/ul
Number of participants experiencing complete response with incomplete count recovery (CRi) from time of transplant to one day following the second treatment | up to 3 months
  Bone marrow aspiration and local peripheral blood counts will be used to measure response. CRi is defined as the following:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of disease, AND
  * Full recovery of peripheral blood counts: platelets > 100,000/ul, and ANC > 1000/ul
Response blast-free hypoplastic or aplastic bone marrow from time of transplant to one day following the second treatment | up to 3 months
  Bone marrow aspiration and local peripheral blood counts will be used to measure response. Blast-free hypoplastic or aplastic bone marrow response is defined as the following:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of disease, AND
  * Full recovery of peripheral blood counts: platelets > 50,000/ul, and ANC > 500/ul
Disease burden measured as the minimal residual disease (MRD) response from time of transplant to one day following the second treatment | up to 3 months
  MRD remission is defined as the occurrence of an MRD level below 10^-4 measured by quantitative reverse transcription polymerase chain reaction (PCR) or flow cytometry.
  Complete response defined as: no detectable leukemic cells by PCR or flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Merin, MD PhD, Principal Investigator — Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States